CLINICAL TRIAL: NCT00711061
Title: Cardiovascular Risk in Growth Hormone Deficient Young Adult Males After Completing Growth Hormone Therapy.
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Carol Huseman, MD, Children's Mercy Hospital
Other Study IDs: 07-07-119E
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 18-25 year old males, growth hormone deficient, who completed growth hormone treatment 3-5 years prior to enrollment in study
- 2: 18-25 year old males, healthy, never treated with growth hormones.

SUMMARY:
The purpose of this study is to compare the cardiovascular risks of growth hormone deficient young adult males who have completed growth hormone therapy to healthy young adult males.

DETAILED DESCRIPTION:
Adults with growth hormone deficiency are at risk for cardiovascular disease. What age this begins is not known.

The objectives of this study are to compare the following measurements between growth hormone deficient young males 3-7 years post completion of growth hormone treatment and age related healthy controls:

1. Carotid artery imaging
2. Metabolic and cardiac parameters
3. Body composition measurements

ELIGIBILITY:
Growth Hormone Deficient Inclusion Criteria:

* Males, 18-25 years old
* Completed growth hormone therapy approximately 3-5 years prior to study enrollment
* History of multiple pituitary hormone deficiencies or growth hormone stimulation test <7 at initiation of growth hormone therapy

Healthy Control Inclusion Criteria:

* Males, 18-25 years old
* No confirmed endocrine diagnosis including Diabetes and thyroid disorders
* BMI - z-score within 2 SD of mean

Exclusion Criteria:

* Known risk factors for cardiovascular disease (eg tobacco use, hypertension, diabetes)
* Family history of early cardiovascular disease (myocardial infarction or stroke <55years of age) in first degree family members
* Any implanted device
* Medication known to interfere with glucose or lipid metabolism or to influence blood pressure
* Chronic organ illness (eg severe asthma, hepatic or nephritic conditions)

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Endocrine clinic and community sample
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Compare carotid artery intima medial thickness | During study visit

SECONDARY OUTCOMES:
Compare metabolic parameters and body composition measurements | During study visit

CONTACTS AND LOCATIONS:
Overall Officials: Carol Huseman, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Childrens Mercy Hospitals and Clinics, Kansas City, Missouri, United States